CLINICAL TRIAL: NCT05888467
Title: The Impact of Physical Activity on the Cardiovascular Profile of Pre-conceptional Women At Risk for Developing Gestational Hypertensive Disorders in Subsequent Pregnancy.
Brief Title: Physical Activity and Cardiovascular Profile of Pre-conceptional Women At Risk for GHD
Acronym: SPORTY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Responsible Party: Principal Investigator, Dr. Dorien Lanssens, Principal Investigator, Hasselt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SPORTY-01
Record Dates: First submitted 2023-05-16; First posted 2023-06-05 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Gestational Hypertension; Cardiovascular Pregnancy Complication
MeSH Terms: conditions — Hypertension, Pregnancy-Induced; Pregnancy Complications, Cardiovascular | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Prospective, monocentric, interventional, randomized-controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control group (Other): non-supervised exercise group
  Interventions: Other: Control group
- Intervention: supervised non-infrared exercise group (Active Comparator): supervised non-infrared exercise group
  Interventions: Other: supervised infrared exercise group
- Intervention: supervised infrared exercise group (Active Comparator): supervised infrared exercise group
  Interventions: Other: supervised non-infrared exercise group

INTERVENTIONS:
Other: supervised infrared exercise group — Participants of the intervention group will be asked to perform 1-3 exercise sessions per week at the Infraligne center of Genk, Hasselt or Maasmechelen for a total duration of 12 weeks. During the exercise session, the participant is assigned to an individual 'sport cabin' in which they are standardly exposed to infrared light.
  Arms: Intervention: supervised non-infrared exercise group
Other: supervised non-infrared exercise group — Participants of the intervention group will be asked to perform 1-3 exercise sessions per week at the Infraligne center of Genk, Hasselt or Maasmechelen for a total duration of 12 weeks. Participants assigned to the supervised non-infrared exercise group will exercise in the sport-cabin with the infrared light turned off.
  Arms: Intervention: supervised infrared exercise group
Other: Control group — Participants of the control group are advised to perform moderate intensity aerobic exercise at least 3 days per week for an average of 30-50 minutes per session and a total duration of 12 weeks.
  Other Names: non-supervised exercise group
  Arms: Control group

SUMMARY:
To compare the cardiovascular profile of pre-conceptional women at risk for developing Gestational Hypertensive Disorders in subsequent pregnancy before and after physical activity.

DETAILED DESCRIPTION:
The SPORTY trial hypothesizes that exercise improves the cardiovascular (CV) profile of pre-conceptional women at risk for developing gestational hypertensive disorders (GHD) in subsequent pregnancy in a profile-specific way.

Research objectives:

The primary objective is to compare the complete CV profile before and after an exercise period of 6 and 12 weeks.

Secondary objectives are:

* To correlate the exercise-induced changes in CV profile to the type, frequency and intensity of exercise.
* To evaluate the added value of supervised and personalized training in inducing changes in the CV profile compared to non-supervised training.
* To evaluate the added value of infrared light therapy during supervised training in inducing changes in the CV profile compared to non-infrared supervised training.
* To assess how long the adaptations in the CV profile induced by supervised training last in case the supervision is halted.

Methodology:

All study participants who provided written informed consent and are eligible to participate in the study are 2:1:1 randomly assigned into a non-supervised exercise group (control), a supervised non-infrared exercise group (intervention), or a supervised infrared exercise group (intervention), stratified by baseline cardiac output (CO).

All study participants will undergo a CV profiling assessment at baseline, at week 6 visit, at week 12 visit, and at week 18 visit. The CV profile assessment is a standardized validated protocol consisting of a simple, non-invasive method using the combination of (1) electrocardiogram (ECG) with Doppler ultrasonography providing information about arteries and veins, (2) Bio-Impedance Spectrum Analysis (BI) using Maltron giving information about the fluid balance, and (3) Impedance Cardiography (ICG) using the NICCOMO registering heart parameters in supine and standing position. The CV profiling will be performed at UHasselt (building A) or at Ziekenhuis Oost-Limburg (Campus Sint-Jan) in the framework of the Limburg Clinical Research Center.

All participants are asked to complete the International Physical Activity Questionnaire (IPAQ) online in Castor EDC at home to report their baseline physical activity status. Demographics, clinical characteristics and medical history are obtained and reported in the eCRF.

For ethical reasons, all study groups will be advised to exercise for a period of 12 weeks, but only the two supervised exercise groups will receive a personalized and guided exercise plan. In addition, all participants will receive an activity diary and are asked to fill in their weekly exercise throughout the entire study period.

ELIGIBILITY:
Inclusion Criteria:

* Women at risk for the development of GHD in subsequent pregnancy based on the presence of at least one of the following risk factors:

  * high body mass index (BMI>30 kg/m²)
  * a family history of PE (mother, sister)
  * in the need of assisted reproduction techniques in a previous or subsequent pregnancy
  * maternal comorbidities: prior PE, diabetes mellitus, chronic hypertension, chronic kidney disease or antiphospholipid syndrome
* Non-pregnant (as confirmed by a negative pregnancy urine dipstick test)
* Age ≥ 18 years
* Being able to understand the Dutch language

Exclusion Criteria:

Participants eligible for this study must not meet any of the following criteria:

* Pregnant at inclusion
* Not being able to exercise according to physician's decision
* Suffering from underlying diseases that can affect the CV profile such as oncological diseases coronary heart disease, aortic disease, peripheral arterial disease
* Participating in another clinical study that may alter the results of this study

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Non-pregnant women at risk for the development of GHD in subsequent pregnancy
Enrollment: 140 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in cardiac output level from Baseline at week 12 visit | Baseline and week 12
  Cardiac Output assessed via the NICCOMO

SECONDARY OUTCOMES:
Change in arterial parameters from Baseline at week 12 visit | Baseline and week 12
  arterial pulse transit time (APTT), pulsatility index (PI) and resistivity index (RI) of the left and right arcuate arteries
Change in venous parameters from Baseline at week 12 visit | Baseline and week 12
  enous pulse transit time (VPTT) of the hepatic and left and right renal veins, hepatic vein impedance index (HVI), and left and right renal interlobar vein impedance indices (RIVI)
Change in cardiac parameters from Baseline at week 12 visit | Baseline and week 12
  stroke volume (SV), systolic blood pressure (SBP), diastolic blood pressure (DBP), mean arterial pressure (MAP), heart rate (HR), pre-ejection period (PEP), total peripheral resistance (TPR), left ventricular ejection time (LVET), velocity and acceleration indices (VI and ACI)
Change in body water volumes from Baseline at week 12 visit | Baseline and week 12
  total body water (TBW), extracellular water (ECW), intracellular water (ICW), ratio ECW/ICW

CONTACTS AND LOCATIONS:
Overall Officials: Dorien Lanssens, Principal Investigator — UHasselt
Locations (1):
- Hasselt University, Diepenbeek, Limburg, Belgium